CLINICAL TRIAL: NCT02707432
Title: Reducing Cardiovascular Disease Risk Factors in Rural Communities in North Carolina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); James McFarlin Community Development, Inc. (Other); Project Momentum, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13-2576; 5R01HL120690-02 (NIH)
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-01

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Community-Based Participatory Research; African Americans
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Permadyne Premier

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time 1 (T1) Intervention Group (Experimental): This group will be the first to receive the adapted intervention, "Heart Matters" (adapted from the PREMIER intervention). The intervention will be 12 months long.
  Interventions: Behavioral: Heart Matters
- Time 2 (T2) Intervention Group (Experimental): This delayed intervention group will receive the adapted intervention, "Heart Matters," six months after the T1 Intervention group. The intervention will be 12 months long.
  Interventions: Behavioral: Heart Matters

INTERVENTIONS:
Behavioral: Heart Matters — "Heart Matters" is an intervention adapted from PREMIER, an evidence-based, comprehensive lifestyle intervention that focuses on blood pressure as the primary outcome. To assess the feasibility and efficacy of adapting PREMIER for rural African Americans, Heart Matters will be delivered to multiple intervention groups, but at two different stages.
  Other Names: PREMIER

SUMMARY:
The study will determine the feasibility and efficacy of adapting an evidence-based intervention (EBI) to reduce cardiovascular disease (CVD) risk factors in rural African American communities and determine the acceptability of mobile technology in these communities to support behavior change.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD), the leading cause of death in the United States (US), disproportionately burdens rural communities. CVD prevalence rates for residents of rural areas (13.1%) is higher compared to those in urban areas (11.2%) of the US. The proposed settings for this research report similar trends in CVD prevalence, where CVD and stroke are among the top three leading causes of death. In community health assessments conducted in the last three years CVD risk factors such as obesity and hypertension were among the top 10 health priorities in our target counties. Compared to residents of metropolitan areas, rural residents have higher rates of cigarette smoking, obesity, mortality from ischemic heart disease, and are physically inactive. These disparities are likely to widen; at the current rate, its estimated 50% of individuals in the US will have CVD by 2030.

Using a community-based participatory research (CBPR) approach, our specific aims for the study are to:

1. Expand and sustain a coalition of community and academic stakeholders to develop successful CVD risk prevention strategies in rural communities;
2. Conduct a mixed-method community needs and assets assessment based on: a) assemble, review and assess existing sources of CVD data; b) identification of community strengths and resources using a web-based survey of community, faith based, social service and healthcare organizations; c) determine the acceptability of components of CVD risk reduction EBIs and community members' perceptions of possible targets for intervention using focus group interviews; d) determine specific family influences (barriers and facilitators) on acceptability of EBI acceptability;
3. Adapt PREMIER, a multi-component EBI using intervention mapping;
4. Conduct a small-scale randomized control trial to assess a) efficacy; and, b) feasibility and adaption of implementing adapted PREMIER in rural settings.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Aged 21 and older
* Has at least one of the following cardiovascular disease (CVD) risk factors: pre-diabetes, hypertension, obesity, family history of early CVD, prior CVD
* Reside in Nash or Edgecombe counties of North Carolina

Exclusion Criteria:

* Evidence of active or unstable CVD
* Cognitive impairment that limits informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Corbie-Smith, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill; Mysha Wynn, MA, Principal Investigator — Project Momentum, Inc.; Shirley McFarlin, BA, Principal Investigator — James McFarlin Community Development, Inc.
Locations (2):
- United States (2):
  - Project Momentum Inc., Rocky Mount, North Carolina
  - Shirley McFarlin, Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frerichs L, Bess K, Young TL, Hoover SM, Calancie L, Wynn M, McFarlin S, Cene CW, Dave G, Corbie-Smith G. A Cluster Randomized Trial of a Community-Based Intervention Among African-American Adults: Effects on Dietary and Physical Activity Outcomes. Prev Sci. 2020 Apr;21(3):344-354. doi: 10.1007/s11121-019-01067-5. PMID 31925605
- [Derived] Corbie-Smith G, Wiley-Cene C, Bess K, Young T, Dave G, Ellis K, Hoover SM, Lin FC, Wynn M, McFarlin S, Ede J. Heart Matters: a study protocol for a community based randomized trial aimed at reducing cardiovascular risk in a rural, African American community. BMC Public Health. 2018 Jul 31;18(1):938. doi: 10.1186/s12889-018-5802-1. PMID 30064398

RESULTS

PARTICIPANT FLOW:
Groups:
- Time 1 Heart Matters Intervention Group: This group will receive the adapted intervention, "Heart Matters" (adapted from the PREMIER intervention) immediately after baseline data collection. Intervention is 26, 90 minute group sessions and 7, 30-60 minute individual sessions across a 1 year period with 1st 6 months intensive period and 2nd 6 months maintenance period.
- Time 2 Heart Matters 6 Month-Delayed Intervention Group: This 6 month delayed intervention group will receive the adapted intervention, "Heart Matters," six months after baseline data collection. Intervention is 26, 90 minute group sessions and 7, 30-60 minute individual sessions across a 1 year period with 1st 6 months intensive period and 2nd 6 months maintenance period.
Period: Overall Study
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group
Started | 72 | 71
Completed | 57 | 51
Not Completed | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group | Total
Number analyzed (Participants) | 72 | 71 | 143
Age, Categorical [Count of Participants; unit: Participants] — Population: Data were available for 139 participants
  Participants
    number analyzed (Participants) | 71 | 68 | 139
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 51 | 40 | 91
    >=65 years | 20 | 28 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data were available for 139 participants
  years
    number analyzed (Participants) | 71 | 68 | 139
    (all) | 54.38 (16.23) | 59.93 (12.64) | 57.26 (14.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data were available for 140 participants
  Participants
    number analyzed (Participants) | 72 | 68 | 140
    Female | 54 | 47 | 101
    Male | 18 | 21 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 71 | 143
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 71 | 143

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Measured in pounds
Time Frame: Baseline and 6 months after initiated treatment
Population: Data reported only for participants with both Baseline and Month 6 data.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group
Number analyzed (Participants) | 37 | 34
pounds | 0.41 (11.23) | 0.92 (10.33)

2. Secondary Outcome: Change in Systolic Blood Pressure
Description: Blood pressure as measured in mmHg
Time Frame: Baseline, Month 6
Population: Data reported only for participants with both Baseline and Month 6 data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group
Number analyzed (Participants) | 38 | 32
mmHg | 8.79 (19.42) | 2.67 (18.01)

3. Secondary Outcome: Change in Diastolic Blood Pressure
Description: As measured in mmHg
Time Frame: Baseline, Month 6
Population: Data reported only for participants with both Baseline and Month 6 data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group
Number analyzed (Participants) | 38 | 32
mmHg | 5.05 (12.96) | 2.00 (10.93)

ADVERSE EVENTS:
Time Frame: From baseline through 18 month follow-up data collection.
Arm/Group | Time 1 Heart Matters Intervention Group | Time 2 Heart Matters 6 Month-Delayed Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/71
Other Adverse Events (participants affected / at risk) | 0/72 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/32/NCT02707432/Prot_SAP_000.pdf